CLINICAL TRIAL: NCT01046136
Title: Double Blind, Randomized, Placebo Controlled Study of Mucinex® for the Treatment of Symptoms of an Acute Respiratory Tract Infection When Two 600 mg Tablets Are Given Every 12 Hours for 7 Days
Brief Title: Mucinex Exploratory Cold Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-MUC-03
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Common Cold
Keywords: common cold
MeSH Terms: conditions — Common Cold | interventions — Guaifenesin; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucinex (Active Comparator)
  Interventions: Drug: guaifenesin (Mucinex)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: guaifenesin (Mucinex) — bid 7 days
  Arms: Mucinex
Drug: placebo — bid 7 days
  Arms: placebo

SUMMARY:
This is an exploratory, multicenter, randomized, blinded, placebo-controlled study of Mucinex in patients with colds. Patients will receive 7 days of treatment with either Mucinex or placebo. The study will assess the effects of Mucinex on sputum and cold symptoms.

ELIGIBILITY:
Inclusion Criteria:

* common cold symptoms
* meet symptom severity
* females of child-bearing potential must have negative pregnancy test and use effective birth control

Exclusion Criteria:

* chronic respiratory conditions
* significant heart, kidney, liver, or lung disease, uncontrolled hypertension or diabetes, cystic fibrosis, thyroid disorder
* pregnant or lactating
* known malignancy
* participation in any other clinical trial within 30 days of baseline
* related to another enrolled patient or persons involved directly or indirectly with the conduct of this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pioneer Clinical Research, Bellevue, Nebraska, United States

REFERENCES:
- [Derived] Hoffer-Schaefer A, Rozycki HJ, Yopp MA, Rubin BK. Guaifenesin has no effect on sputum volume or sputum properties in adolescents and adults with acute respiratory tract infections. Respir Care. 2014 May;59(5):631-6. doi: 10.4187/respcare.02640. Epub 2013 Sep 3. PMID 24003241
- [Derived] Albrecht H, Vernon M, Solomon G. Patient-reported outcomes to assess the efficacy of extended-release guaifenesin for the treatment of acute respiratory tract infection symptoms. Respir Res. 2012 Dec 27;13(1):118. doi: 10.1186/1465-9921-13-118. PMID 23270519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from waiting rooms of health care providers/clinics between December 2009 and March 2010.
Pre-assignment Details: Participants screened over 2 day period who suffer from an acute respiratory tract infection.
Groups:
- Mucinex: 2 X 600 MG TABLETS EVERY 12 HOURS FOR 7 DAYS
- Placebo: 2 TABLETS EVERY 12 HOURS FOR 7 DAYS
Period: Overall Study
Arm/Group | Mucinex | Placebo
Started | 188 | 190
Completed | 184 | 182
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mucinex | Placebo | Total
Number analyzed (Participants) | 188 | 190 | 378
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 6
  Between 18 and 65 years | 178 | 175 | 353
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.91) | 40.8 (15.04) | 41.0 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 84 | 180
  Male | 92 | 106 | 198
Region of Enrollment [Number; unit: participants]
  United States | 188 | 190 | 378

OUTCOME MEASURES:

1. Primary Outcome: Investigator's End of Study Assessment of Treatment
Description: Yes the investigator would use this treatment for cold symptoms in the future.
Time Frame: 7 days
Population: MITT defined as all participants receiving at least 1 dose of study medication and had 1 or more efficacy assessment after Baseline. Last observation carried forward method was applied to missing post baseline measurement in the analyses of the MITT population.
Measure: Number; unit: participants
Groups:
- Mucinex: Two 600mg tablets taken taken twice daily
- Placebo: Two placebo tablets, identical in appearance to active treatment, taken taken twice daily
Arm/Group | Mucinex | Placebo
Number analyzed (Participants) | 178 | 180
participants | 163 | 149
Statistical Analysis 1: Comparison: Mucinex vs Placebo; Investigator's End-of-Study Assessment NOTE: All assessments of efficacy were considered exploratory and were given equal consideration, and were carried out on both the MITT and PP populations. LOCF method was applied to missing post baseline measurements in analyses of the MITT population; Test type: Superiority or Other; p = 0.0096, Regression, Logistic; p-value is from a logistic regression model with terms for treatment group and center

2. Secondary Outcome: Number of Patients With Adverse Events
Description: Total number of patients with adverse events that were possibly or probably related.
Time Frame: 7 days
Population: All participants who received study medication, excluding participants who later returned all the dispensed study medication to the site unused.
Measure: Number; unit: participants
Arm/Group | Mucinex | Placebo
Number analyzed (Participants) | 188 | 189
participants | 12 | 6

3. Primary Outcome: Mean Change From Baseline in a 6 Point Severity Scale (0 = None, 1 = Very Mild, 2 = Mild or Slight, 3 = Moderate, 4 = Severe or 5 = As Bad as it Can be) for Cough.
Description: Mean change from baseline in a 6 point severity scale between treatment groups(0 = None, 1 = Very mild, 2 = Mild or slight, 3 = Moderate, 4 = Severe or 5 = As bad as it can be) for cough.
Time Frame: Baseline and Day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mucinex | Placebo
Number analyzed (Participants) | 183 | 186
units on a scale | -1.1 (0.14) | -0.9 (0.14)
Statistical Analysis 1: Comparison: Mucinex vs Placebo; Test type: Superiority or Other; p = 0.0293, Wilcoxon (Mann-Whitney); P-value is from a Wilcoxon rank sum test comparing the two treatment groups

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the treatment period. All patients who received at least 1 dose of study medication were included in the safety analysis.
Arm/Group | Mucinex | Placebo
Serious Adverse Events (participants affected / at risk) | 1/188 | 0/189
Other Adverse Events (participants affected / at risk) | 0/188 | 0/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex (N=188) | Placebo (N=189)
arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) — SAE considered not related to study medication. All SAEs in this study were for one patient and related to one event that occurred 17 days prior to treatment start date.
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) — SAE considered not related to study medication. All SAEs in this study were for one patient and related to one event that occurred 17 days prior to treatment start date.
Lymphatic duct injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — SAE considered not related to study medication. All SAEs in this study were for one patient and related to one event that occurred 17 days prior to treatment start date.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — SAE considered not related to study medication. All SAEs in this study were for one patient and related to one event that occurred 17 days prior to treatment start date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less